CLINICAL TRIAL: NCT05916248
Title: Clinical Study of Personalized Tumor Vaccines mRNA-0217/S001 and Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: Combination Therapy of Personalized mRNA-0217 Vaccines and Pembrolizumab in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Xinpu BioTechnology Company Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021PCV001
Record Dates: First submitted 2023-06-02; First posted 2023-06-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor
Keywords: Personalized neoantigen tumor vaccine; PD-1 inhibitor
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: This clinical trial adopts Bayesian optimal interval (BOIN) design method to determine the maximum tolerated dose (MTD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoantigen tumor vaccine and pembrolizumab combination arm (Experimental): Dose Escalation Phase vaccine: 0.2mg, 0.4mg, 1mg Dose Expansion Phase vaccine : MTD or 1mg Pembrolizumab: 200mg/dose
  Interventions: Biological: Personalized neoantigen tumor vaccine; Biological: PD-1 inhibitor
- Neoantigen tumor vaccine monotherapy arm (Experimental): Dose Escalation Phase vaccine: 0.2mg, 0.4mg, 1mg Dose Expansion Phase vaccine : MTD or 1mg
  Interventions: Biological: Personalized neoantigen tumor vaccine

INTERVENTIONS:
Biological: Personalized neoantigen tumor vaccine — Neoantigen tumor vaccine
Biological: PD-1 inhibitor — pembrolizumab
  Arms: Neoantigen tumor vaccine and pembrolizumab combination arm

SUMMARY:
The main objective of this study was to observe and evaluate the safety and tolerability of mRNA-0217/S001 vaccine encoding personalized tumor neoantigens alone/in combination with Pembrolizumab injection for the treatment of advanced solid tumors. The secondary objective was to observe the preliminary efficacy of mRNA-0217/S001 personalized tumor vaccine in the treatment of advanced solid tumors with neoantigen-specific CD4+ and CD8+ T lymphocyte responses, objective tumor response rate (ORR) and disease control rate (DCR), progression-free survival (PFS) and overall survival (OS) caused by mRNA-0217/S001 personalized tumor vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed written informed consent files,Able to comply with the study protocol, in the investigator's judgment
2. Subjects must be >/= 18 years of age at time of informed consent, regardless of gender
3. Subjects with locally advanced, recurrent or metastatic solid tumors confirmed by histology or cytology within the past 6 months, who have failed standard treatment or are currently not suitable for standard treatment
4. No copy number variations (CNVs) or loss of heterozygosity (Loss-of heterozygosity, LOH) were found in HLA-related genes and chromosomal regions by gene sequencing
5. Advanced or metastatic lesions confirmed by immunohistochemistry, and cryopreserved tissues/cells, enough for WES and RNAseq sequencing, and predicted by bioinformatics analysis, at least one antigen effectively presented by self-HLA was found , such as KRAS or TP53 mutations and correspondingly presented HLA types
6. Life expectancy ≥ 4 months
7. Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
8. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
9. Have adequate organ and bone marrow function,No use of granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), red blood cell transfusion and platelet transfusion within 14 days before the examination
10. Fertile eligible patients (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) during the trial and at least 90 days after the last dose. female patients of childbearing age before the first dose A blood pregnancy test within 7 days must be negative
11. Subjects need to undergo virological examination: those without CMV and EBV, HIV, HBV, HCV, and syphilis infection (only in the baseline period)

Exclusion Criteria:

1. Has had chemotherapy, hormone therapy, traditional Chinese medicine with antitumor indications, or other antitumor therapies deemed to conflict with the current treatment by the investigator within 4 weeks prior to the first administration of the study drug
2. Subjects have undergone major surgical procedures other than the diagnosis or biopsy of the current tumor within 4 weeks before the first dose of mRNA-0217/S001, or are expected to undergo major surgery during the study period
3. Subjects have received allogeneic hematopoietic stem cell transplantation or organ transplantation in the past, or those who plan to receive organ transplantation during this study
4. Subjects have previously received other tumor vaccines or cell therapy
5. Brain metastases with clinical symptoms, spinal cord compression, cancerous meningitis, or other evidence that the brain and spinal cord metastases have not been controlled, and the researchers judged that they are not suitable for enrollment
6. Other malignant tumors known to be progressing or requiring active treatment in the past 2 years (except for non-melanoma skin cancer, superficial bladder cancer, and carcinoma in situ of the cervix that have been cured by surgical curative treatment)
7. History of interstitial lung disease (ILD), pulmonary fibrosis
8. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to a) severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrioventricular block corrected QTc interval male > 450 milliseconds, female > 470 milliseconds, b) Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration, c) New York Heart Association (NYHA) ≥ III heart failure or left ventricular ejection fraction (LVEF) < 50%
9. Other serious and/or uncontrollable diseases, which may affect the subject's participation in this study, include but not limited to a) a history of severe drug allergy, or is known to be allergic to any tumor vaccine and pembrolizumab formulation components or has had severe allergic reactions to other monoclonal antibodies in the past, b) A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, c) Evidence of severe or uncontrolled liver or kidney disease, d) Uncontrolled high blood pressure, diabetes, etc., e) Patients with active ulcers, gastrointestinal bleeding, f) Serious infection requiring intravenous antibiotics or hospitalization or uncontrolled active infection within 4 weeks before the first dose, g) have an active syphilis infection
10. Participate in other clinical trials within 4 weeks before the first dose (except for screening failure)
11. Those who are currently receiving systemic steroids (except those who have recently or currently used inhaled steroids)
12. Pregnant and lactating women
13. Imaging (CT or MRI) shows that the tumor invades large blood vessels and has a tendency to hemorrhage
14. Have clinically significant thyroid dysfunction, and the investigator judges that they are not suitable for enrollment
15. Active pneumonia found in chest CT scan during the screening period
16. Uncontrolled pleural effusion, pericardial effusion, or ascites that needs repeated drainage
17. Subjects who have adverse reactions of the previous anti-tumor therapy have not recovered to NCI-CTCAE 5.0 grade evaluation ≤ grade 1 (except for hair loss)
18. HBsAg positive and peripheral blood HBV DNA detection value is higher than the upper limit of normal, and/or HCV Ab positive and HCV RNA detection value is higher than the upper limit of normal
19. Researchers believe that there are other reasons that are not suitable for participating in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or Dose-limiting toxicity(DLT) | Day1 to Day21
Percentage of Participants With Adverse Events (AEs) | Up to 54 weeks
  Percentage of Participants with Adverse Events (AEs) by Severity According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Biologically Effective Dose (BED). | Day1 to Day21
  if MTD is not reached, BED will be used.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 54 weeks
  Progression-free Survival of Personalized mRNA Tumor Vaccine
overall survival (OS) | Up to 54 weeks
  Overall Survival of Personalized mRNA Tumor Vaccine
Reaction of antigen-specific T cells in peripheral blood | Up to 54 weeks
  mRNA-0217/S001 personalized tumor vaccine induced neoantigen-specific CD4+ and CD8+ T lymphocyte responses
Objective response rate (ORR) | Up to 54 weeks
  ORR calculates the ratio of the number of patients whose best response is complete remission (CR) or partial remission (PR) to the total number of evaluable patients according to RECIST 1.1 criteria. Those who have not been evaluated for lesion and tumor response will be regarded as non-evaluable patients and will not be counted.
disease control rate (DCR) | Up to 54 weeks
  DCR calculates the ratio of the number of patients whose best response is complete remission (CR), or partial remission (PR), or stable disease (SD) to the total number of evaluable patients according to RECIST 1.1 criteria. Those who have not been evaluated for lesion and tumor response will be regarded as non-evaluable patients and will not be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, M.D.&Ph.D, Study Director — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No